CLINICAL TRIAL: NCT03639129
Title: Improving Characterization of Calcifications With Contrast-Enhanced Mammography
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201709088
Record Dates: First submitted 2018-07-31; First posted 2018-08-20 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Mammography
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Contrast-enhanced mammography (CME) (Experimental): -Patients who meet eligibility criteria and consent to participate in this study will complete a CEM examination prior to or on the day that biopsy is scheduled. CEM must occur no later than 60 days after the diagnostic mammogram. The standard of care biopsy must occur no later than 30 days after CEM.
  Interventions: Device: Contrast-enhanced mammography; Procedure: Biopsy

INTERVENTIONS:
Device: Contrast-enhanced mammography — Contrast-enhanced mammography was FDA approved in 2012 and is currently being used in both clinical and research settings at breast imaging centers throughout the world
  Other Names: CME
Procedure: Biopsy — Standard of care

SUMMARY:
The purpose of this study protocol is to assess whether contrast-enhanced mammography (CEM) will increase the accuracy of characterization of microcalcifications detected on screening mammography prior to biopsy as either benign, high risk, or malignant.

ELIGIBILITY:
Inclusion Criteria:

* Women with calcifications detected on screening mammogram for which biopsy is recommended following characterization on diagnostic mammography.
* At least 30 years of age.
* Able to understand and willing to sign an IRB-approved written informed consent document
* GFR ≥ 30 mL/min/1.73 m2

Exclusion Criteria:

* Pregnant
* Prior history of allergy or hypersensitivity reaction to iodinated contrast
* History of chronic renal disease (including dialysis, kidney transplant, single kidney, renal cancer, or renal surgery)
* Patients with known thyroid disorders, pheochromocytoma or sickle cell anemia

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-31 (Estimated); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate risk characterization of screen-detected calcifications by CEM | Up to 30 days after the CEM
  -The proportion of women with abnormal enhancement (yes/no) will be compared to the pathology results from the core needle biopsy (benign versus high risk/malignant)

SECONDARY OUTCOMES:
Rate of detection of additional sites of disease in the same or contralateral breast on CEM | At the time of the CEM (day 1)
  This will be defined as presence of abnormal enhancement in the same breast at least 2 cm away from the margin of the calcifications of interest or any presence of abnormal enhancement in the contralateral breast at the time of CEM
  -The reference standard in this case will also be based on pathology results from core needle biopsy (if additional biopsies are performed) or findings on surgical pathology if the patient elects for mastectomy, with the decision for core needle biopsy and lumpectomy vs mastectomy according to surgeon preference and standard of care.
Ability of CEM to determine whether accuracy for cancer detection varies as a function of breast density | At the time of the CEM (day 1)
  -Breast density category is routinely reported in the screening mammography report and accepted categories include predominantly fatty, scattered fibroglandular densities, heterogeneously dense, and extremely dense.
Ability of whether CEM accuracy for cancer detection varies as a function of the morphology of calcifications as depicted on screening and diagnostic mammography | At the time of the CEM (day 1)
  -Morphology of calcifications include amorphous, coarse heterogeneous, fine pleomorphic, or fine linear branching and/or based on distribution of the calcifications as either diffuse, regional, grouped, linear, or segmental, according to the descriptors in the imaging reports

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Covington, M.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu